CLINICAL TRIAL: NCT05499312
Title: Efficacy and Safety of an Innovative Chinese Herbal Formula for the Treatment of Gout: A Double-blind, Randomized, Placebo-Controlled Trial
Brief Title: An Innovative Chinese Herbal Formula for the Treatment of Gout
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gout Study
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HKIIM-KU formula (Experimental): Subjects will receive HKIIM-KU formula granules (16.9g twice daily) for 8 weeks.
  Interventions: Drug: HKIIM-KU formula
- Placebo (Placebo Comparator): Subjects will receive placebo granules (16.9g twice daily) for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HKIIM-KU formula — Subjects will receive HKIIM-KU formula granules (16.9g twice daily) for 8 weeks.
  Other Names: HKIIM-KU
  Arms: HKIIM-KU formula
Drug: Placebo — Subjects will receive placebo granules (16.9g twice daily) for 8 weeks.
  Arms: Placebo

SUMMARY:
Gout is a chronic disease of deposition of monosodium urate crystals, which form in the presence of increased urate concentrations. Gout is closely related to hyperuricaemia. Urate deposits in the joint, causing joint swelling, pain, movement disorders, affecting a significant portion of the population worldwide annually.

The underlying pathophysiology of gout is multifactorial, complex, and poorly understood. Thus, gout remains one of the major therapeutic challenges. Currently, western medicine treatment of gout flare includes colchicine, NSAIDs and glucocorticoids. These drugs act as analgesics, anti-inflammatory and uric acid lowering drugs. Besides, management of gout and prevention of acute flares of gout make a crucial part in gout management. To obtain uricemia target, urate lowering treatment (ULT) has been widely used in conventional management of gout. Allopurinol, probenecid and febuxostat are some of the examples of ULT. Although researchers have carried out various studies on this disease, there are severe side effects for patients with gout. Therefore, it is necessary to explore new treatments for gout with good efficacy and less side effects.

Chinese medicine (CM) is nowadays widely used for managing gout in China and other East Asian countries. Our principal Investigator (Prof. Zhi-xiu Lin), a highly experienced Registered Chinese Medicine Practitioner working at the School of Chinese Medicine, The Chinese University of Hong Kong, has been using a herbal formula (HKIIM-KU formula) to treat patients with gout in Hong Kong for many years. This formula has been observed to be effective in relieving and preventing gout and its related clinical manifestations. Hence, a double-blind, randomized, placebo-controlled, multicenter clinical trial will be employed in this study, and it would be able to provide robust clinical evidence on the efficacy and safety of HKIIM-KU formula for gout.

DETAILED DESCRIPTION:
Gout is a chronic disease of deposition of monosodium urate crystals, which form in the presence of increased urate concentrations. Gout is closely related to hyperuricaemia. Urate deposits in the joint, causing joint swelling, pain, movement disorders. Gout affects a significant portion of the population worldwide annually. According to a recent meta-analysis, the prevalence of gout world-wide is 0.6%, while there was marked statistical heterogeneity geographically resulting of a prevalence ranging from <1% to 6.8%. The frequent attack of gout not only seriously affect the life of patients, but also lead to disability.

There are a few disease states of gout including asymptomatic hyperuricaemia, acute gouty arthritis, intercritical period, and chronic gouty arthritis. Acute flare of gout is characterized by inflamed joint arthritis which peaks within hours with signs of inflammation including redness, hotness, tenderness, swelling and loss of function. The acute attack usually resolves in 2 weeks and the patient enter into a remission phase called intercritical period. There are usually no symptoms during this period, however, proper treatment for hyperuricaemia is needed to prevent further acute attack of gout. Untreated gout or hyperuricaemia will progress into destruction of joints with formation of tophi which are accumulated monosodium urate (MSU) crystals. Joint destruction and deformity are the untreated results of gout, leading to great distress and disability.

The underlying pathophysiology of gout is multifactorial, complex, and poorly understood. It has been found that environment, genetics, immunity, diet, internal environment, trauma and stimulation are involved in the pathogenesis in various degrees. Thus, gout remains one of the major therapeutic challenges. Currently, western medicine treatment of gout flare includes colchicine, NSAIDs and glucocorticoids. These drugs act as analgesics, anti-inflammatory and uric acid lowering drugs. The mechanism of these drugs is to reduce joint inflammation, pain and uric acid level. Besides, management of gout and prevention of acute flares of gout make a crucial part in gout management. To obtain uricemia target, urate lowering treatment (ULT) has been widely used in conventional management of gout. Allopurinol, probenecid and febuxostat are some of the examples of ULT. Although researchers have carried out various studies on this disease, there are severe side effects for patients with gout. For example, Benzbromarone may cause severe renal damage. Moreover, various studies have found a strong association between human leukocyte antigen-B*58:01 (HLA-B*58:01) and allopurinol-induced severe cutaneous adverse reactions especially in Han Chinese. With such genetic predisposition, patients may develop toxic epidermal necrolysis, Steven Johnson syndrome and other life-threatening immune-mediated severe cutaneous adverse reactions with allopurinol use. It is reported that the carrier rate of the HLA-B*58:01 allele was 14% in Han Chinese in Hong Kong. Therefore, it is necessary to explore new treatments for gout with good efficacy and less side effects.

Chinese medicine (CM) is nowadays widely used for managing gout in China and other East Asian countries. In Traditional Chinese medicine (TCM), gout is classified as Bi pattern usually due to Qi stagnation in the meridians and collaterals. Among them, Zhu Liangchun Gout Decoction is one of the most commonly used formulae. Our principal Investigator (Prof. Zhi-xiu Lin), a highly experienced Registered Chinese Medicine Practitioner working at the School of Chinese Medicine, The Chinese University of Hong Kong, has been using a herbal formula (HKIIM-KU formula) to treat patients with gout in Hong Kong for many years. The formula was based on Zhu Liangchun Gout Decoction and has been modified to suit gout patients in Hong Kong. This formula has been observed to be effective in relieving and preventing gout and its related clinical manifestations. Hence, a double-blind, randomized, placebo-controlled, multicenter clinical trial will be employed in this study, and it would be able to provide robust clinical evidence on the efficacy and safety of HKIIM-KU formula for gout.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meeting the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2015 gout classification criteria (met sufficient criterion* or total score ≥8) ;
2. History of >=1 self-reported flare of gouty arthritis within 12 months prior to randomization;
3. Agree to undergo blood test and willing to complete questionnaires and take medications as scheduled; and
4. Agree to participate in the study and provide written informed consent. (for those illiterate subjects, their family member can sign the consent form upon subject's agreement) Note: * Sufficient criterion = Presence of MSU crystals in a symptomatic joint or bursa (i.e., in synovial fluid) or tophus

Exclusion Criteria:

1. Liver-kidney yin deficiency pattern according to Chinese medicine theory;
2. Use of urate-lowering drugs within 2 weeks prior to screening;
3. Present of tophi or known history of kidney stones.
4. Known use of oral/injectable corticosteroids or other Chinese herbal medicine for treating gout within 1 month prior to screening;
5. Ongoing acute gout arthritis flare at screening or within 2 weeks prior to screening;
6. History of >4 flares overall in the 12 months prior to screening.
7. Polyarticular gouty arthritis involving more than 4 joints;
8. Severe deformity, stiffness and labor loss of patients with advanced arthritis;
9. Known rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis;
10. Known history of any serious diseases such as severe kidney and liver impairments, autoimmune disease, thyroid disease, Hodgkin's disease, lymphoma, severe mental disorders and leukemia
11. Known presence or suspicion of acute infectious disease;
12. Known history of malignancy within the past 5 years;
13. Known allergic to the drug used in this study;
14. Documented pregnant or lactation;
15. Subjects participating in other clinical studies at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Serum uric acid | week 4
  Blood sample for serum uric acid (sUA) will be collected. It is regarded as a controllable factor that contributing to gout. Evidence showed that gout flare risk increases when a patient's sUA fails to achieve target level.
Serum uric acid | week 8
  Blood sample for serum uric acid (sUA) will be collected. It is regarded as a controllable factor that contributing to gout. Evidence showed that gout flare risk increases when a patient's sUA fails to achieve target level.

SECONDARY OUTCOMES:
Serum uric acid | week 12
  Blood sample for serum uric acid (sUA) will be collected. It is regarded as a controllable factor that contributing to gout. Evidence showed that gout flare risk increases when a patient's sUA fails to achieve target level.
Pain Visual Analogue Scale | week 2
  Pain VAS is validated for assessing chronic gout. A 0-10 point visual analog scale is used to reflect the pain the patient had due to gout in the past week, where score of 0 and 10 representing "No pain" and "Severe pain" respectively.
Pain Visual Analogue Scale | week 4
  Pain VAS is validated for assessing chronic gout. A 0-10 point visual analog scale is used to reflect the pain the patient had due to gout in the past week, where score of 0 and 10 representing "No pain" and "Severe pain" respectively.
Pain Visual Analogue Scale | week 8
  Pain VAS is validated for assessing chronic gout. A 0-10 point visual analog scale is used to reflect the pain the patient had due to gout in the past week, where score of 0 and 10 representing "No pain" and "Severe pain" respectively.
Pain Visual Analogue Scale | week 12
  Pain VAS is validated for assessing chronic gout. A 0-10 point visual analog scale is used to reflect the pain the patient had due to gout in the past week, where score of 0 and 10 representing "No pain" and "Severe pain" respectively.
Health Assessment Questionnaire Disability Index | week 2
  HAQ-DI is a validated tool for measuring physical function in patients with gout.
Health Assessment Questionnaire Disability Index | week 4
  HAQ-DI is a validated tool for measuring physical function in patients with gout.
Health Assessment Questionnaire Disability Index | week 8
  HAQ-DI is a validated tool for measuring physical function in patients with gout.
Health Assessment Questionnaire Disability Index | week 12
  HAQ-DI is a validated tool for measuring physical function in patients with gout.
Short Form-36 | week 2
  Short Form-36 is a validated tool to assess health-related quality of life in patients with gout. It has been proven to be responsive to change in gout especially its physical component summary.
Short Form-36 | week 4
  Short Form-36 is a validated tool to assess health-related quality of life in patients with gout. It has been proven to be responsive to change in gout especially its physical component summary.
Short Form-36 | week 8
  Short Form-36 is a validated tool to assess health-related quality of life in patients with gout. It has been proven to be responsive to change in gout especially its physical component summary.
Short Form-36 | week 12
  Short Form-36 is a validated tool to assess health-related quality of life in patients with gout. It has been proven to be responsive to change in gout especially its physical component summary.
No. of patients with new flare | Up to week 12
  Number of patients with at least one new gout flare after baseline
Time to first new flare | Up to week 12
  Time to the first new gout flare
Number of patients using rescue medication | Up to week 12
  Number of patients using rescue medication (i.e. paracetamol) after baseline
Time to first use of rescue medication | Up to week 12
  Time to first use of rescue medication after baseline
Adverse events | Up to week 12
  Adverse events related to study treatment will be recorded.
Clinical pattern/syndrome according to Chinese medicine theory | Up to week 12
  Subjects will be assessed by Registered Chinese Medicine Practitioners (RCMPs) under Chinese medicine theory in this trial. A form will be used to record the clinical pattern/syndrome on each visit by the RCMP according to Chinese medicine theory.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu LIN, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong